CLINICAL TRIAL: NCT02254421
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Multi-Center Study Evaluating Antiviral Effects, Pharmacokinetics, Safety, and Tolerability of GS-5806 in Hematopoietic Cell Transplant (HCT) Recipients With Respiratory Syncytial Virus (RSV) Infection of the Lower Respiratory Tract
Brief Title: Presatovir in Hematopoietic Cell Transplant Recipients With Respiratory Syncytial Virus (RSV) Infection of the Lower Respiratory Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-218-1502; 2014-002475-29 (EudraCT Number)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Respiratory Syncytial Virus (RSV); Antiviral; Hematopoietic Cell Transplant (HCT); Lower respiratory tract infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — presatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Presatovir (Experimental): Participants will receive presatovir on Days 1, 5, 9, 13, and 17, with follow-up visits through Day 28, and may continue in an optional extended monitoring phase with visits through Day 56.
  Interventions: Drug: Presatovir
- Placebo (Placebo Comparator): Participants will receive placebo to match presatovir on Days 1, 5, 9, 13, and 17, with follow-up visits through Day 28, and may continue in an optional extended monitoring phase with visits through Day 56.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Presatovir — Presatovir 200 mg (4 × 50 mg tablets) administered orally or via nasogastric (NG) tube
  Other Names: GS-5806
  Arms: Presatovir
Drug: Placebo — Placebo to match presatovir administered orally or via nasogastric tube
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of presatovir on respiratory syncytial virus (RSV) viral load in autologous or allogeneic hematopoietic cell transplant (HCT) recipients with an acute RSV lower respiratory tract infection (LRTI).

ELIGIBILITY:
Key Inclusion Criteria:

* Received an autologous or allogeneic HCT using any conditioning regimen
* Evidence of new abnormalities on chest X-ray obtained < 48 hours prior to screening, determined to be consistent with LRTI by the local radiologist, relative to the most recent previous chest X-ray. If chest X-ray is not available, a chest X-ray must be obtained for screening.
* Documented RSV in both the upper (eg, nasal swab, nasopharyngeal swab, nasal wash) and lower (eg, induced sputum, bronchoalveolar lavage, lung biopsy, but not spontaneous sputum) respiratory tract as determined by local testing (eg, polymerase chain reaction, direct fluorescence antibody, respiratory viral panel assay, or culture). All samples must have been collected ≤ 6 days prior to Day 1, or as determined at screening as per protocol.
* An informed consent document signed and dated by the participant or a legal guardian of the participant and investigator or his/her designee.
* A negative urine or serum pregnancy test is required for female participants (unless surgically sterile or greater than two years post-menopausal)
* Male and female participants of childbearing potential must agree to contraceptive requirements as described in the study protocol
* Willingness to complete necessary study procedures and have available a working telephone or email

Key Exclusion Criteria:

Related to concomitant or previous medication use:

* Use of non-marketed (according to region) investigational agents within 30 days, OR use of any monoclonal anti-RSV antibodies within 4 months or 5 half-lives of screening, whichever is longer, OR use of any investigational RSV vaccines after HCT
* Use of a moderate or strong cytochrome P450 enzyme inducer including but not limited to rifampin, St. John's Wort, carbamazepine, phenytoin, efavirenz, bosentan, etravirine, modafinil, and nafcillin, within 2 weeks prior to the first dose of study drug

Related to medical history:

* Pregnant, breastfeeding, or lactating females
* Unable to tolerate nasal sampling required for this study, as determined by the investigator
* Known history of HIV/AIDS with a CD4 count <200 cells/μL within the last month
* History of drug and/or alcohol abuse that, in the opinion of the investigator, may prevent adherence to study activities

Related to medical conditions:

* Requiring invasive mechanical ventilation at the time of randomization
* Documented to be positive for other respiratory viruses (limited to influenza, parainfluenza, human rhinovirus, adenovirus, human metapneumovirus, or coronavirus), from the lower respiratory tract sample as determined by local testing
* Clinically significant bacteremia or fungemia within 7 days prior to screening that has not been adequately treated, as determined by the investigator
* Clinically significant bacterial, fungal, or viral pneumonia within 2 weeks prior to screening that has not been adequately treated, as determined by the investigator
* Excessive nausea/vomiting at screening, as determined by the investigator, or an inability to swallow pills that precludes oral administration of the investigational medical product (for individuals without an NG tube in place)
* Any condition which, in the opinion of the investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints

Related to laboratory results:

* Creatinine clearance < 30 mL/min (calculated using the Cockcroft-Gault method)
* Clinically significant aspartate aminotransferase/alanine aminotransferase, as determined by the investigator
* Clinically significant total bilirubin, as determined by the investigator

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (17):
- United States (11):
  - City of Hope, Duarte, California
  - University of Chicago, Chicago, Illinois
  - John Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - New York Weill Cornell Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchison Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - Hopital Saint-Louis, APHP, Paris
  - Hopital Foch, Suresnes
  - CHU de Bordeaux, Talence
- Seoul Saint Mary's Hospital, Seoul, South Korea
- Karolinska Institutet, Stockholm, Sweden
- University Clinical Basel, Basel, Switzerland

REFERENCES:
- [Derived] Marty FM, Chemaly RF, Mullane KM, Lee DG, Hirsch HH, Small CB, Bergeron A, Shoham S, Ljungman P, Waghmare A, Blanchard E, Kim YJ, McKevitt M, Porter DP, Jordan R, Guo Y, German P, Boeckh M, Watkins TR, Chien JW, Dadwal SS. A Phase 2b, Randomized, Double-blind, Placebo-Controlled Multicenter Study Evaluating Antiviral Effects, Pharmacokinetics, Safety, and Tolerability of Presatovir in Hematopoietic Cell Transplant Recipients with Respiratory Syncytial Virus Infection of the Lower Respiratory Tract. Clin Infect Dis. 2020 Dec 31;71(11):2787-2795. doi: 10.1093/cid/ciz1167. PMID 31915807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia Pacific, Europe, and the United States. The first participant was screened on 31 January 2015. The last study visit occurred on 17 April 2017.
Pre-assignment Details: 71 participants were screened.
Groups:
- Presatovir: Presatovir 200 mg (4 x 50 mg tablets) on Days 1, 5, 9, 13, and 17 administered orally or via nasogastric tube
- Placebo: Placebo tablets on Days 1, 5, 9, 13, and 17 administered orally or via nasogastric tube
Period: Overall Study
Arm/Group | Presatovir | Placebo
Started | 31 | 29
Completed | 29 | 26
Not Completed | 2 | 3
Not completed — Randomized but Not Treated | 1 | 0
Not completed — Death | 0 | 2
Not completed — Withdrew Consent | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 full dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Presatovir | Placebo | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (16.27) | 54.4 (12.59) | 52.4 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 21 | 23 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 3 | 7
  Black or African American | 1 | 2 | 3
  White | 23 | 18 | 41
  Not Permitted | 1 | 5 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 23 | 18 | 41
  Not Permitted | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 2 | 2 | 4
  Sweden | 0 | 1 | 1
  United States | 27 | 20 | 47
  France | 1 | 3 | 4
  Switzerland | 0 | 3 | 3
Stratification Factor: Supplemental O2 Requirement at Time of Randomization [Count of Participants; unit: Participants]
  Supplemental O2 Requirement ≤ 2 L/min | 19 | 19 | 38
  Supplemental O2 Requirement > 2 L/min | 11 | 10 | 21
Stratification Factor: Treatment of Current RSV Infection with Ribavirin [Count of Participants; unit: Participants]
  Yes | 12 | 11 | 23
  No | 18 | 18 | 36
Nasal Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] | 6.22 (1.365) | 6.02 (1.574) | 6.12 (1.462)
Oxygen Saturation [Mean (Standard Deviation); unit: percent saturation] — Oxygen saturation is a measure of how much oxygen the blood is carrying as a percentage of the maximum it could carry.
  percent saturation | 94 (3.8) | 93 (5.1) | 93 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average Change in Nasal Respiratory Syncytial Viral (RSV) Load From Baseline to Day 9
Description: The time-weighted average change, often referred to as the DAVG, provides the average viral burden change from baseline. The mean values presented were calculated using the ANCOVA model and are adjusted for baseline value and stratification factors.
Time Frame: Baseline to Day 9
Population: Full Analysis Set: all randomized participants who received at least 1 full dose of study drug and had an RSV viral load greater than or equal to the lower limit of quantification of the RT-qPCR assay in the Day 1 nasal sample, as determined by RT-qPCR at the central lab.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 29 | 28
log10 copies/mL | -1.00 (0.215) | -0.97 (0.218)
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.94, ANCOVA — P-value was calculated from the ANCOVA model including baseline values and stratification factors; Treatment difference = -0.02, 95% CI 2-sided [-0.62 to 0.57]

2. Secondary Outcome: Number of Supplemental O2-Free Days Through Day 28
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 29 | 28
days | 26 [10 to 28] | 28 [9 to 28]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.84, Negative binomial — P-value was calculated from the negative binomial model with stratification factors as covariates

3. Secondary Outcome: Percentage of Participants Developing Respiratory Failure Requiring Mechanical Ventilation Through Day 28
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 29 | 28
percentage of participants | 10.3 [2.2 to 27.4] | 10.7 [2.3 to 28.2]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.98, Cochran-Mantel-Haenszel — P-value was calculated from the Cochran-Mantel-Haenszel (CMH) test stratified by stratification factors

4. Secondary Outcome: Percentage of All-Cause Mortality Among Participants Through Day 28
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Presatovir | Placebo
Number analyzed (Participants) | 29 | 28
percentage of participants | 0.0 [0.0 to 11.9] | 7.1 [0.9 to 23.5]
Statistical Analysis 1: Comparison: Presatovir vs Placebo; Test type: Superiority; p = 0.19, Cochran-Mantel-Haenszel — P-value was calculated from the CMH test stratified by stratification factors

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: Safety Analysis Set: participants who received at least 1 full dose of study drug.
Arm/Group | Presatovir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 4/29
Serious Adverse Events (participants affected / at risk) | 7/30 | 7/29
Other Adverse Events (participants affected / at risk) | 19/30 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=30) | Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Graft versus host disease (Immune system disorders) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Presatovir (N=30) | Placebo (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2
Visual impairment (Eye disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 3
Acute sinusitis (Infections and infestations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Troponin T increased (Investigations) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (8):
  • Study Protocol: Original (2014-06-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_008.pdf
  • Study Protocol: Amendment 1 (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_009.pdf
  • Study Protocol: Amendment 2 (2014-09-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_010.pdf
  • Study Protocol: Amendment 3 (2014-10-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_011.pdf
  • Study Protocol: Amendment 5 (Amendment 4 not implemented) (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_012.pdf
  • Study Protocol: Amendment 6 (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_013.pdf
  • Study Protocol: Amendment 7 (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/Prot_014.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02254421/SAP_015.pdf